CLINICAL TRIAL: NCT05403333
Title: Weekly Utidelone in HER2-negative Inoperable Locally Advanced or Metastatic Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Chief Physician, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DOUBLE
Record Dates: First submitted 2022-04-18; First posted 2022-06-03 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-05

CONDITIONS: Breast Neoplasms; Locally Advanced or Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Utidelone (Experimental): Drug: utidelone Utidelone Injection: 65 mg/m2/day, IV on day 1, 8, and 15 every 28 days
  Interventions: Drug: utidelone

INTERVENTIONS:
Drug: utidelone — Utidelone Injection: 65 mg/m2/day, IV on day 1, 8, and 15 every 28 days
  Other Names: Singel arm

SUMMARY:
This is a phase II trial to explore the efficacy and safety of weekly utidelone in HER2-negative inoperable locally advanced or metastatic breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent Form;
* Women aged ≥ 18 years;
* Histologically or cytologically confirmed HER2-negative locally advanced or metastatic breast cancer:

  * The most recent pathology confirmed HER2 negative, defined as HER2 0/1 + by standard immunohistochemical staining (IHC) or HER2 2 + by IHC but negative by in situ hybridization (ISH);
  * Patients with locally advanced or locally recurrent disease should be unable to undergo radical surgical resection confirmed by the investigators;
* Eastern Cooperative Oncology Group (ECOG) score [0-2] points;
* At least one evaluable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST1.1):

  * If there is only bone metastasis, it is required that the bone metastasis lesion contains bone destruction component;
  * if there is only pleural effusion, it is required that the pleural effusion is malignant confirmed by pathology
* No more than 2 prior lines of chemotherapy for advanced and/or metastatic disease;
* Prior chemotherapy regimens must have included taxane;
* Patients with hormone receptor positive disease received at least one line of endocrine therapy for metastatic disease (including CDK4/6 inhibitors, everolimus, chidamide and PI3K inhibitors, etc.);
* Patients must have recovered to ≤ Grade 1 (CTCAE v5.0) from all toxicities related to prior anticancer therapy. with the following exceptions: 1). alopecia; 2). pigmentation;
* Adequate hematological, hepatic and renal function;
* Life expectancy of at least 12 weeks;
* Patients must be able to participate and comply with treatment and follow-up.

Exclusion Criteria:

* Previous treatment with UTD-1;
* Patients with other malignant tumors within 5 years prior to enrollment, except cured cutaneous basal cell carcinoma and cervical carcinoma in situ;
* Anti-tumor therapy, including chemotherapy, radical radiotherapy, biological therapy, immunotherapy or anti-tumor Chinese medicine therapy within 4 weeks prior to the start of study treatment; endocrine therapy within 2 weeks prior to the start of study treatment;
* Patients who have undergone major organ surgery (excluding needle biopsy) or have significant trauma within 4 weeks prior to study treatment, or need to undergo elective surgery during the trial;
* Patients with clinically suspected brain metastases. However, patients who have received previous treatment for central nervous system metastasis (radiotherapy or surgery) can be included if they have been confirmed as stable by imaging for at least 4 weeks and have stopped symptomatic treatment (including hormone and mannitol, etc.) for more than 2 weeks;
* Patients with active HBV, HCV and HIV infection; except patients with stable hepatitis B after drug treatment (DNA titer should not be higher than 500 IU/mL or copy number < 1000 copies/ml) and patients with cured hepatitis C (HCV RNA test negative);
* Peripheral neuropathy ≥grade 2 (CTCAE 5.0) and patients with grade 1 peripheral neuropathy will be enrolled at the discretion of the investigator;
* Prior grade 3 or above nervous system-related adverse events caused by previous use of anti-microtubule drugs;
* Pregnant or lactating female patients or fertile women with positive baseline pregnancy test; or subjects of childbearing potential who are unwilling to take effective contraceptive measures during the study period and within at least 90 days after the last dose;
* Known or suspected hypersensitivity to any of the study drugs or excipients;
* Exclusion of any other non-malignant systemic diseases (cardiovascular, renal, hepatic, etc.) that preclude the implementation or follow-up of the treatment regimen; • Any other condition that the investigator considers inappropriate for participation in this trial.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2022-06-10 (Estimated); Primary Completion 2023-03-09 (Estimated); Study Completion 2025-03-09 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | Estimated 12 months
  PFS is defined as the duration from enrollment to the first radiologically confirmed progressive disease (PD) (RECIST 1.1 criteria) or death due to any cause.

SECONDARY OUTCOMES:
Objective response rate (ORR) | Estimated 12 months
  The proportion of patients with a best response of CR or PR, according to RECIST 1.1 criteria
Overall Survival (OS) | Estimated 24 months
  From enrollment to death (for any reason)
Duration of Response (DOR) | Estimated 12 months
  The first evaluation of CR or PR to progression or death (for any reason)
Overall summary of adverse events following intravenous administration of utidelone (safety analysis set) | Estimated 12 months
  Incidence of treatment-emergent adverse events based the Common Terminology Criteria for Adverse Events (CTCAE) version 5.0[ Time Frame: 1 years] Observe and record incidence of adverse events and severe adverse events associated with utidelone treatment, assessed by investigators according to CTCAE version 5.0.

IPD SHARING:
Plan to Share IPD: Undecided